CLINICAL TRIAL: NCT03853759
Title: COMPARİSON OF HEART FAİLURE PATİENTS AND HEALTHY PEOPLE İN BALANCE AND GAİT PARAMETERS
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, E.Burcu ÖZCAN, COMPARİSON OF HEART FAİLURE PATİENTS AND HEALTHY PEOPLE İN BALANCE AND GAİT PARAMETERS, Hacettepe University
Other Study IDs: GO 18/736-06
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure,Balance
Keywords: Gait Parameters, Heart Failure,Balance,Gait,Cognition,Functional Capacity,Muscle Strength
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Heart Failure
- Healthy İndividuals

SUMMARY:
We aimed to show the difference between balance and gait parameters in heart failure and healthy individuals.

DETAILED DESCRIPTION:
Heart failure is the inability of the heart to pump a sufficient amount of blood into our body. The reason is usually the decrease in the contractile capacity of myocardium due to decreased coronary blood flow. Symptoms and symptoms may be quite diverse in the underlying pathophysiology of heart failure, which is usually the only type. As a result of heart failure; problems such as dyspnoea, anemia, peripheral edema, peripheral muscle involvement and decreased muscle mass, confusion, sleep disorder, dementia, various cardiac symptoms and renal failure can be seen.

Balance body with minimal muscle activity in static or dynamic position on the support base is to maintain the center of gravity. Patients with heart failure may have decreased postural control, exercise intolerance, breathing problems, and decreased cognitive function.

Gait analysis, evaluation of neuro musculoskeletal system functions and interpretation of results with numbers and graphs. Gait analysis is an analysis method that plays a role in many cases of clinical diagnosis and follow-up. Heart failure is characterized by a significant reduction in walking distance, which leads to reduced quality of life. In a study conducted in heart failure, it is stated that gait velocity is a determinant of one year mortality and hospitalization, and should be considered for clinical evaluations and prognosis. All these causes of heart failure in chronic disease groups defined considering it is important to investigate the balance and gait parameters.

This study will show the difference between the balance and walking parameters in heart failure according to the healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction <40% or less,
* Without acute decompensation,
* No revascularization in the last six months,
* The drug has been stable for the last four weeks,
* Accepts participation in the study,
* Coopere,
* NewYork Heart Association -NYHA Class II- III
* Patients with heart failure who are amputated without support or assistive devices will be included in the study.

Exclusion Criteria:

* Neurological, cognitive or orthopedic diseases that affect the measurements,
* Severe respiratory disease (FEV1 <35%),
* BNP> 100pg / ml and above,
* Acute infection,
* Resting heart rate above 140 beats / min,
* Dementia,
* Having a BMI> 35 or above,
* Individuals with other chronic diseases that may affect their balance and walking will not be included in the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: İndividuals who are diagnosed with Heart Failure at Hacettepe University and who reffered to the Cardiopulmonary Rehabilitation Unit for Physiotherapy also who are willing to participate in the study will be include in the study.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Balance Assesment | 1st Day
  Balance Assesment will be evaluated with Mini-Balance Evaluation Systems Test (Mini-BESTest) The Mini-BESTest includes four subscales: transitions/anticipatory postural control, reactive postural control, sensory orientation and stability in gait. Each item is rated on a three-point ordinal scale (0 = severe to 2 = normal). t the MiniBESTest consists of 14 items, with a maximum score of 28 points. The Mini-BESTest takes 10 to 15 minutes to administer.
Gait Parameters | 1st Day
  Gait Parameters assesment using Biodex Gait Trainer It will be evaluated from the basic walking parameters in terms of walking speed, double step length, number of steps per minute, step cycle and ambulation index.

SECONDARY OUTCOMES:
Cognition | 1st Day
  Cognition Using Mini Mental State Examination Test (MMSE) Cognitive function will be evaluated the screening tool the Mini Mental State Examination (MMSE)
Exercise Capacity | 1st Day
  Exercise Capacity Using 6-Minute Walk Test The standard protocol of the test is applied in a 30 meter continuous corridor.Standard instructions are given during testing.
Muscle Strength | 1st Day
  Muscle Strength assesment M.Quadriceps Femoris muscles strength will be evaluated non-invasive methods by measuring muscle dynamometer device. Both legs will be measured.
Level of Physical Activity | 1st Day
  Level of Physical Activity Assesment Using The International Physical Activity Questionnaires (IPAQ) The questionnaire consists of seven questions and provides information on the time spent in walking, mid-severe activities
Balance Confidence | 1st Day
  Balance Confidence Using Activity Specific Balance Confidence Scale (ABC) This scale contains 16 tasks related to indoor and outdoor daily living activities

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes